CLINICAL TRIAL: NCT01519583
Title: Title: Comparative Effectiveness of Pedometer-Based Walking Interventions: WalkMore
Brief Title: WalkMore Walking Interventions for Overweight/Obese Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 11018
Record Dates: First submitted 2012-01-18; First posted 2012-01-27 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Postmenopausal Disorder; Blood Pressure; Over Weight
Keywords: walking; physical activity; sedentary behavior
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Basic Pedometry Intervention (Experimental): Basic pedometry intervention: Participants will have a goal of obtaining 10,000 steps/day (with no direction with regards to walking intensity/speed/cadence)
  Interventions: Behavioral: Basic Intervention
- Enhanced Pedometry Intervention (Experimental): Enhanced pedometry Intervention: Participants will have the goal of obtaining 10,000 steps/day and at least 30 minutes in moderate intensity (i.e., at a cadence of at least 100 steps/min);
  Interventions: Behavioral: Enhanced Pedometry
- Control Group (Placebo Comparator): Control group: Will maintain their usual activity and return for follow-up measures
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Basic Intervention — Participants will have the goal of obtaining 10,000 steps/day. In addition, participants will attend a meeting once a week with study staff, during which pedometers will be checked, and staff will provide a behavioral intervention to improve physical activity levels
  Other Names: Pedometry
  Arms: Basic Pedometry Intervention
Behavioral: Enhanced Pedometry — Intensity Enhanced Pedometry: Participants will have the goal of obtaining 10,000 steps/day at least 30 minutes in moderate intensity (i.e., at a cadence of at least 100 steps/min). In addition, participants will attend a meeting once a week with study staff, during which pedometers will be checked, and the staff will provide a behavioral intervention to improve physical activity levels.
  Arms: Enhanced Pedometry Intervention
Behavioral: Control Group — Maintain usual physical activity, and return for follow-up measures.
  Other Names: No Pedometry
  Arms: Control Group

SUMMARY:
The WalkMore study will help find out how walking interventions can help overweight/obese postmenopausal women with increased risk of cardiovascular disease lower their blood pressure.

DETAILED DESCRIPTION:
Baseline assessment, then a three month intervention or control condition, followed by another assessment at the end of the study. Participants will be screened for blood pressure, height, weight, and the distance around the waist. Participants who meet the eligibility criteria will be given a pedometer to log steps for one week. During visit 2, participants will return the pedometer, and are able to self-monitor appropriately, they will be given an accelerometer to wear for one week.

Pedometry:

Participants will wear a small device which will measure the amount of steps accumulated for 7 days during the first week of the run-in period and again at follow-up (Control group will not perform follow-up pedometry).

Accelerometry:

Participants will be asked to wear a small device similar to a pedometer attached to a belt at the hip to measure physical activity levels for 7 days during the second week of the run-in period and again at the week prior to follow-up.

Assessment Visits (Baseline and 3 Months):

Blood pressure, brachial ultrasound (measure of the health of the artery), blood draw (fasting blood glucose and insulin), height, body weight, and waist measurement will be measured at the beginning of the main study and again after the 3-month period.

Brachial Artery Ultrasound:

An ultrasound is a procedure that uses sound waves to create a picture. The brachial artery ultrasound measures how elastic the arteries are and the thickness of the lining of the major blood vessel in the upper arm (the brachial artery). After resting for fifteen minutes, an ultrasound probe will be placed over the brachial artery in the elbow area on the non-dominant arm. A blood pressure cuff will be inflated around the forearm for five minutes to reduce blood flow. When the cuff is deflated, the ultrasound will be continued for five more minutes to observe the blood flowing back into the arm.

Blood Draw:

A fasting blood draw will occur to obtain fasting glucose and insulin.

Walking Gait:

Participants will walk across a 16 foot computerized floor mat, which will measure walking speed. After a couple practice walks, the participant will be asked to walk 2 times across the mat at 6 different self-selected paces: very slow, slow, preferred/normal, fast, very fast, and as quickly as possible (without running). The participant will be able to rest as needed. The computerized mat will measure walking speed and other elements associated with the pace at which the participant walks.

ELIGIBILITY:
Inclusion Criteria:

* Woman between 45-74 years of age
* Have not had a menstrual period for at least 12 months
* Are not regularly physically active (self-reported non-exerciser for previous 6 months)
* Have a body mass index (BMI) between 25-45 kg/m2
* Have high normal blood pressure or (systolic pressure of 130-179 mmHg or a diastolic pressure of 85-99 mmHg)
* Not limited in your ability to walk
* Understand these criteria
* Are willing to provide informed consent
* Willing to be randomized to either type of walking intervention or a control group being studied, and are willing to follow the protocol for the group to which they have been assigned

Exclusion Criteria:

* Have a past history and/or physical examination or laboratory findings of a medical condition including (but not limited to):
* Have any medical condition or disease that is life-threatening or that can interfere with or be aggravated by exercise
* Have been diagnosed with diabetes
* Blood pressure is greater than 179 mmHg systolic or 99 mmHg diastolic.
* Participating in another research study which may effect the results of WalkMore

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Resting systolic blood pressure | 3 Months
  Measured in the seated position using AHA blood pressure measurement guidelines

SECONDARY OUTCOMES:
Resting diastolic blood pressure | 3 Months
  Diastolic blood pressure is measured in the seated position in accordance with AHA guidelines
Accelerometry | 3 Months
  An Accelerometry is a device that measures the amount of physical activity.
Brachial Ultrasound | 3 Months
  Brachial Ultrasound is a measurement of the health of the artery, which measures the ability of the brachial artery to dilate.
Waist Circumference | 3 Months
  Waist Circumference is the distance measured around the waist
Walking gait | 3 Months
  Walking gait is evaluated through the use of an electronic mat, which measures walking speed and other elements of gait.

CONTACTS AND LOCATIONS:
Overall Officials: Catrine Tudor-Locke, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Tudor-Locke C, Schuna JM, Swift DL, Dragg AT, Davis AB, Martin CK, Johnson WD, Church TS. Evaluation of Step-Counting Interventions Differing on Intensity Messages. J Phys Act Health. 2020 Jan 1;17(1):21-28. doi: 10.1123/jpah.2018-0439. PMID 31698336
- [Derived] Tudor-Locke C, Swift DL, Schuna JM Jr, Dragg AT, Davis AB, Martin CK, Johnson WD, Church TS. WalkMore: a randomized controlled trial of pedometer-based interventions differing on intensity messages. BMC Public Health. 2014 Feb 15;14:168. doi: 10.1186/1471-2458-14-168. PMID 24528783